CLINICAL TRIAL: NCT03292978
Title: Probiotics Intervention on Gut Flora Metabolisms of Choline:A Randomized Double-Blind Control Trial
Brief Title: An Intervention on Healthy Adults of Probiotics on Gut Flora Metabolisms of Choline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huilian Zhu (Other)
Responsible Party: Sponsor-Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DIC2016-08
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics intervention (Experimental): 1. The probiotic is provided in sachets as a 2g powder dried with corn starch.
  2. The powder is orally taken once daily for 4 weeks.
  3. The powder contains totally 11 log 10 colony forming units(CFU) of probiotics.
  4. The types of probiotics are Lactobacillus.rhamnosus, Lactobacillus.acidophilus, Bifidobacteria.animalis and Bifidobacteria.longum.
  Interventions: Dietary Supplement: probiotics intervention
- non-probiotic control (Placebo Comparator): The placebo is corn starch alone provided and the shape, color, weight,flavor and taste are same with the powder of probiotics intervention.
  Interventions: Dietary Supplement: non-probiotic control

INTERVENTIONS:
Dietary Supplement: probiotics intervention — The probiotics intention is provided with 4 strains of probiotics as a 2g sachet powder, dried with corn starch for 4 weeks.
  Arms: probiotics intervention
Dietary Supplement: non-probiotic control — The placebo is corn starch alone provided and the shape, color, flavor and taste are same with the powder of probiotics intervention.
  Arms: non-probiotic control

SUMMARY:
The aim of the study is to examine the effects of probiotics intervention on choline metabolites and intestinal microbiota composition using a randomized double blind clinical trial. Also, we proposed to explore the real-time change of choline metabolites after probiotics intervention through a PC challenge test. Our study will clarify the biochemical pathway involved in metabolic diseases and hope to provide a new targeted-preventive and therapeutic strategy for chronic metabolic diseases.

DETAILED DESCRIPTION:
Dietary choline (mainly refer to phosphatidylcholine, PC) produce trimethylamine (TMA) through the action of gut flora in vivo. TMA then readily absorbed into systemic circulation and oxidized by hepatic flavin monoxygenases (FMO3) to trimethylamine-N-oxide (TMAO). The elevated levels of circulating TMAO is identified as a risk factor for the prevalence and development of metabolic diseases such as cardiovascular diseases and nonalcoholic fatty liver diseases. Targeting gut flora for reducing TMAO may be a promising approach for preventing chronic metabolic diseases. Recent studies found that some strains representing two different phyla (Firmicutes and Proteobacteria) are capable of producing TMA from choline in vitro. On the other hand, TMA intervention can change the structure of intestinal flora, reducing the abundance of bifidobacterium and lactobacillus. Probiotics can improve the ecological balance of the gut flora, which might be beneficial to human health and disease prevention. However, whether probiotics could inhibit the TMA-producing bacterias and reduce the TMA and TMAO levels through balancing the gut flora was unclear.

In order to explore whether probiotics can reduce the TMA and TMAO levels, we are proposed to recruit 50 volunteers aged from 18-30 years old to participate in the randomized double-blind trial. The volunteers are randomized allocated into different intervention groups. The probiotics intervention group is provided once daily orally-taken powder in a sachet, which contains 4 strains of probiotics. The non-probiotic control is provided with a powder without probiotics , but has same look, color, taste, flavor and weight as the probiotics intervention group. A PC challenge test will be hold before and after the 4 weeks intervention. The blood and fecal sample will be collected before and after the trial and analyzed by appropriate method. The dietary assessment is assessed by a 3-day dietary record.The statistic analysis is by SPSS 23.0.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males at 18 to 30 years old;
* Free from antibiotics and probiotic products for at least 1 month;
* Willing to participate in the study, consume the test product and perform all measurements.

Exclusion Criteria:

* Sever physical diseases;
* Intolerance to probiotics or eggs

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
choline metabolites | 4 weeks later
  The metabolites of choline before and after the intervention including free choline, betaine, TMA, TMAO will be measured by UPLC/MS.

SECONDARY OUTCOMES:
intestinal microbiota composition | 4 weeks later
  The intestinal microbiota composition of feces before and after the intervention will be examined by 16S-DNA.
anthropometry measurement | 4 weeks later
  The height and weight which are combined to report BMI in kg/m^2 will be measured before and after the intervention by professional investigators.
blood biochemical markers | 4 weeks later
  Overnight fasting serum total cholesterol (TC), triglyceride (TG), LDL cholesterol (LDLc), HDL cholesterol (HDLc) and fasting blood glucose were measured by colorimetric methods using a Hitachi 7600-010 automated analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Hui lian, Professor, Study Chair — Sun Yat-sen University
Locations (1):
- SunYat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen S, Jiang PP, Yu D, Liao GC, Wu SL, Fang AP, Chen PY, Wang XY, Luo Y, Long JA, Zhong RH, Liu ZY, Li CL, Zhang DM, Zhu HL. Effects of probiotic supplementation on serum trimethylamine-N-oxide level and gut microbiota composition in young males: a double-blinded randomized controlled trial. Eur J Nutr. 2021 Mar;60(2):747-758. doi: 10.1007/s00394-020-02278-1. Epub 2020 May 21. PMID 32440731